CLINICAL TRIAL: NCT04664413
Title: Correlations Between Percentage of BRAFV600E Alleles and Outcome in Thyroid Carcinoma
Brief Title: Percentage of BRAFV600E Alleles and Outcome in Thyroid Carcinoma
Acronym: ABOUT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Salerno (Other)
Responsible Party: Principal Investigator, Mario Vitale, professor, University of Salerno
Other Study IDs: ABOUT
Record Dates: First submitted 2020-12-05; First posted 2020-12-11 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Papillary Thyroid Cancer
MeSH Terms: conditions — Thyroid Cancer, Papillary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 3 adjacent slides of formalin-fixed, paraffin-embedded (FFPE) tissues. One devoted to microscopy analysis; two for DNA and RNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
BRAFV600E is the most frequent oncogene in Papillary thyroid carcinoma (PTC). It correlates with greater extension, lymph node metastasis, and advanced stage. However, the prognostic value of BRAFV600Eis weak and the search of this mutation is not recommended in clinical management of thyroid cancer.

PTC are characterized by intratumor heterogeneity with wild-type and BRAFV600E tumoral cells. In a previous study, the BRAFV600E/BRAFwild-type ratio correlated with patient age, tumor volume, lymph node metastasis and with worst disease outcome. While the existence of intratumor heterogeneity in PTC is supported by many evidences, its extension, biological signiﬁcance and clinical utility is questioned and must be further investigated.

Primary endpoint of the study is to determine the relationship between the percentage of BRAFV600E alleles and outcome in PTC patients. Secondary endpoints are to determine the mean and median BRAFV600E/BRAFwild-type allele ratio in heterogeneous tumors; determine the relationship between the percentage of BRAFV600E alleles and clinicopathological features.

The study protocol entails the assessment by digital-droplet PCR the BRAFV600E/BRAFwild-type allele ratio in a series of PTC and its correlation with clinicopathology features and outcome.

DETAILED DESCRIPTION:
BACKGROUND Papillary thyroid carcinoma (PTC) generally shows an excellent prognosis with a 5-year survival of over 95%. Even when PTC metastasizes to the regional lymph nodes, a frequent occurrence, it generally has an excellent prognosis. However, there are some patients who present with an aggressive background or with specific clinicopathological features who exhibit aggressive developmental behavior. Several clinicopathological features, namely pathology subtype, age, distant and lymph node metastasis, extrathyroid extension, and completeness of resection can be used to predict prognosis and have been adopted in staging systems such as the AMES, MACIS, and AJCC TNM classifications.

The genetic background is a powerful prognostic determinant only when applied to some gene mutations such as TERT promoter and p53 mutations. The prognostic value of BRAFV600E, the most frequent oncogene in PTC, is weak. It correlates with greater extension, lymph node metastasis, and advanced stage (III/IV). Its correlation with outcome in PTC has been the object of many not always concordant studies. A large multicenter study was necessary to unequivocally demonstrate the association between BRAFV600E and cancer recurrence and mortality. The risk of PTC harboring BRAFV600E remains weak (recurrence hazard ratio 2.66) and the search of this mutation is not recommended in clinical management of low-risk patients with thyroid cancer.

Different research groups provided evidence on the heterogeneity of PTC that consist of a mixture of tumor cells with wild-type and BRAFV600E (5, 6). The importance of the percentage of BRAFV600E positive cells within the tumor was demonstrated in 168 PTC. The analysis of BRAFV600E/BRAFwild-type ratio was performed by pyrosequencing and higher ratio positively correlated with patient age, tumor volume, lymph node metastasis and with worst disease outcome. Patients with tumors with BRAFV600E/BRAFwild-type ratio ≥ 30% displayed an odds risk of tumor recurrence of 5.1, whereas it was only 1.75 in BRAFV600E positive tumors if the allele ratio was not considered. The qualitative analysis BRAFV600E positive versus negative PTC can explain the discordant correlations with clinicopathological features and outcome in different cohorts of patients with different ratio of BRAFV600E alleles, and ultimately the qualitative analysis BRAF mutational status can reduce the strength of its clinical significance and utility.

While the existence of intratumor heterogeneity in PTC is supported by many evidences, its extension, biological signiﬁcance and clinical utility is questioned and must be further investigated.

Digital-droplet PCR (ddPCR) is an analytical method recently developed, suitable for absolute quantification of target DNA in a DNA mixture. It is the most accurate method to determine the BRAFV600E/BRAFwild-type allele ratio.

AIM OF THE RESEARCH

1. Determine how frequent are subclonal-BRAFV600E PTC and to determine the mean and median BRAFV600E/BRAFwild-type allele ratio in heterogeneous tumors;
2. Determine the relationship between the percentage of BRAFV600E alleles and clinicopathological features;
3. Determine the relationship between the percentage of BRAFV600E alleles and outcome in PTC patients (primary endpoint)

STUDY DESIGN

* A large series of PTC formalin-fixed, paraffin-embedded (FFPE) tissues with a clinical follow up > 3 years will be analyzed by ddPCR to determine the percentage of BRAFV600E alleles.
* The purity of PTC samples and the ratio neoplastic cell/contaminating cells will be assessed by the a) analysis by rt-PCR of expression of a panel of RNA specific for lymphoreticular cells and stromal cells; b) microscopic review of adjoining tissue sections.
* Statistical analysis will be performed to search correlations between percentage of BRAFV600E alleles and a) pathology features, TNM, staging; b) recurrence and survival

ELIGIBILITY:
Inclusion Criteria:

* Patients undergone surgery because of any PTC subtypes 3 years before or more
* Availability of PTC tissue samples, well annotated
* Availability of clinical data of the patients including gender, age at diagnosis, type and extension of surgery, radiation therapy, radio-iodide therapy, TSH suppressive therapy
* Follow up of 3 years or more after surgery, including periodical 6 months assessment of TSH, thyroglobulin and AbTG, neck ultrasound evaluation and episodic hrTSH stimulation test

Exclusion Criteria:

* Inadequate tissue samples or clinical data and follow up
* Purity of PTC samples < 50%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient 18 years age or more with a diagnosis of papillary thyroid carcinoma, subjected to thyroidectomy no less than 3 years before
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Intratumor BRAFV600E heterogeneity and outcome | 6 months
  3. Determine the relationship between the percentage of BRAFV600E alleles and outcome in PTC patients

SECONDARY OUTCOMES:
Intratumor BRAFV600E heterogeneity quantification | 5 months
  1. Determine how frequent are subclonal-BRAFV600E PTC and to determine the mean and median BRAFV600E/BRAFwild-type allele ratio in heterogeneous tumors
Intratumor BRAFV600E heterogeneity and clinicopathological features | 5 months
  2. Determine the relationship between the percentage of BRAFV600E alleles and clinicopathological features

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine and Surgery, Univeristy of Salerno, Baronissi, Salerno, Italy

IPD SHARING:
Plan to Share IPD: Undecided
All results, will be shared before any submission to scientific journal

REFERENCES:
- [Background] Ito Y, Miyauchi A, Kihara M, Fukushima M, Higashiyama T, Miya A. Overall Survival of Papillary Thyroid Carcinoma Patients: A Single-Institution Long-Term Follow-Up of 5897 Patients. World J Surg. 2018 Mar;42(3):615-622. doi: 10.1007/s00268-018-4479-z. PMID 29349484
- [Background] Xing M, Westra WH, Tufano RP, Cohen Y, Rosenbaum E, Rhoden KJ, Carson KA, Vasko V, Larin A, Tallini G, Tolaney S, Holt EH, Hui P, Umbricht CB, Basaria S, Ewertz M, Tufaro AP, Califano JA, Ringel MD, Zeiger MA, Sidransky D, Ladenson PW. BRAF mutation predicts a poorer clinical prognosis for papillary thyroid cancer. J Clin Endocrinol Metab. 2005 Dec;90(12):6373-9. doi: 10.1210/jc.2005-0987. Epub 2005 Sep 20. PMID 16174717
- [Background] Xing M, Alzahrani AS, Carson KA, Shong YK, Kim TY, Viola D, Elisei R, Bendlova B, Yip L, Mian C, Vianello F, Tuttle RM, Robenshtok E, Fagin JA, Puxeddu E, Fugazzola L, Czarniecka A, Jarzab B, O'Neill CJ, Sywak MS, Lam AK, Riesco-Eizaguirre G, Santisteban P, Nakayama H, Clifton-Bligh R, Tallini G, Holt EH, Sykorova V. Association between BRAF V600E mutation and recurrence of papillary thyroid cancer. J Clin Oncol. 2015 Jan 1;33(1):42-50. doi: 10.1200/JCO.2014.56.8253. Epub 2014 Oct 20. PMID 25332244
- [Background] Xing M, Alzahrani AS, Carson KA, Viola D, Elisei R, Bendlova B, Yip L, Mian C, Vianello F, Tuttle RM, Robenshtok E, Fagin JA, Puxeddu E, Fugazzola L, Czarniecka A, Jarzab B, O'Neill CJ, Sywak MS, Lam AK, Riesco-Eizaguirre G, Santisteban P, Nakayama H, Tufano RP, Pai SI, Zeiger MA, Westra WH, Clark DP, Clifton-Bligh R, Sidransky D, Ladenson PW, Sykorova V. Association between BRAF V600E mutation and mortality in patients with papillary thyroid cancer. JAMA. 2013 Apr 10;309(14):1493-501. doi: 10.1001/jama.2013.3190. PMID 23571588
- [Background] Guerra A, Sapio MR, Marotta V, Campanile E, Rossi S, Forno I, Fugazzola L, Budillon A, Moccia T, Fenzi G, Vitale M. The primary occurrence of BRAF(V600E) is a rare clonal event in papillary thyroid carcinoma. J Clin Endocrinol Metab. 2012 Feb;97(2):517-24. doi: 10.1210/jc.2011-0618. Epub 2011 Dec 14. PMID 22170714
- [Background] Gandolfi G, Sancisi V, Torricelli F, Ragazzi M, Frasoldati A, Piana S, Ciarrocchi A. Allele percentage of the BRAF V600E mutation in papillary thyroid carcinomas and corresponding lymph node metastases: no evidence for a role in tumor progression. J Clin Endocrinol Metab. 2013 May;98(5):E934-42. doi: 10.1210/jc.2012-3930. Epub 2013 Mar 26. PMID 23533235
- [Background] Guerra A, Fugazzola L, Marotta V, Cirillo M, Rossi S, Cirello V, Forno I, Moccia T, Budillon A, Vitale M. A high percentage of BRAFV600E alleles in papillary thyroid carcinoma predicts a poorer outcome. J Clin Endocrinol Metab. 2012 Jul;97(7):2333-40. doi: 10.1210/jc.2011-3106. Epub 2012 Apr 16. PMID 22508706